CLINICAL TRIAL: NCT06621849
Title: The Effect of Unilateral Erector Spinae Plane Block Versus Intrathecal Morphine on Early Mobilization After Total Hip Replacement Under Spinal Anesthesia in Cairo University Hospitals: a Prospective Randomized Clinical Study
Brief Title: Effect of Unilateral Erector Spinae Plane Block Versus Intrathecal Morphine on Early Mobilization After Hip Replacement
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim Hussein, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-259-2024
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
Keywords: erector spinae plane block, morphine, hip replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group {E} (Experimental): patients in this group will receive Erector spinae plane block on the ipsilateral side of the surgery then 3.5 ml of bupivacaine 0.5% and 0.25 ml of normal saline intrathecal
  Interventions: Procedure: erector spinae plane block
- Group {M} (Active Comparator): patients in this group will receive 5 ml of subcutaneous lidocaine 1% then 3.5 ml of bupivacaine 0.5% and 0.1 mg of morphine in 0.25 ml of normal saline intrathecal.
  Interventions: Drug: Morphine

INTERVENTIONS:
Procedure: erector spinae plane block — In the erector spinae plane block (group E), an ultrasound-guided block will be performed on the ipsilateral side of the surgery while the patient is in lateral position 3-5 cm from the midline (10). Moving cephalic from the sacrum, we will identify the L5, L4, and L3 transverse processes and erector spinae muscles posteriorly. A 21 G and 70mm length needle will be directed in-plane, and the needle tip will be positioned anterior to the erector spinae muscle at the corner of the transverse process. After the initial saline injection, dissection of the plane will be observed by injecting a total volume of 20 ml composed of 10 micrograms dexmedetomidine in 2ml of normal saline and 18 ml of bupivacaine 0.25%, which is far from the toxic dose (10). Correct placement is defined as the spread of local anesthetic cranially and caudally from the injection point, dissecting the plane between the transverse processes and erector spinae muscles.
  Arms: Group {E}
Drug: Morphine — patients will receive 5 ml of subcutaneous lidocaine 1% then 3.5 ml of bupivacaine 0.5% and 0.1 mg of morphine in 0.25 ml of normal saline intrathecal
  Other Names: oramorph
  Arms: Group {M}

SUMMARY:
* Preoperative assessment: Patients who fulfill inclusion criteria will be evaluated by medical history, physical examination and clinical laboratory tests which are a complete blood picture (CBC), kidney function tests, liver function tests, international normalized ratio(INR), prothrombin time(PT), and chest X-Ray. An electrocardiograph (ECG) will be done for patients above 40 years old. Patients will be prepared by 8 hours of preoperative fasting, receiving a tablet of Omeprazole 20 mg and Alprazolam 0.5 mg at bedtime the day before surgery.
* All patients will be educated about the standard Numerical Rating Scale (NRS) for pain score of 0-10 (0 = no pain, 10 = the most severe pain) during preanesthetic evaluation visit.
* In our study, 70 patients will be randomly divided into two equal groups, with 35 pt. in each. Spinal anesthesia will be performed at L3-L4 with 3.5 ml of hyper¬baric bupivacaine 0.5% and 0.25 ml normal saline only for the E group or 0.1 mg morphine in 0.25 ml normal saline for the M group (9).

Group {E} will receive ESPB on the ipsilateral side of the surgery then 3.5 ml of bupivacaine 0.5% and 0.25 ml of normal saline intrathecal.

Group {M} will receive 5 ml of subcutaneous lidocaine 1% then 3.5 ml of bupivacaine 0.5% and 0.1 mg of morphine in 0.25 ml of normal saline intrathecal.

DETAILED DESCRIPTION:
* Preoperative assessment: Patients who fulfill inclusion criteria will be evaluated by medical history, physical examination and clinical laboratory tests which are a complete blood picture (CBC), kidney function tests, liver function tests, international normalized ratio(INR), prothrombin time(PT), and chest X-Ray. An electrocardiograph (ECG) will be done for patients above 40 years old. Patients will be prepared by 8 hours of preoperative fasting, receiving a tablet of Omeprazole 20 mg and Alprazolam 0.5 mg at bedtime the day before surgery.
* All patients will be educated about the standard Numerical Rating Scale (NRS) for pain score of 0-10 (0 = no pain, 10 = the most severe pain) during preanesthetic evaluation visit.
* In our study, 70 patients will be randomly divided into two equal groups, with 35 pt. in each. Spinal anesthesia will be performed at L3-L4 with 3.5 ml of hyper¬baric bupivacaine 0.5% and 0.25 ml normal saline only for the E group or 0.1 mg morphine in 0.25 ml normal saline for the M group (9).

Group {E} will receive ESPB on the ipsilateral side of the surgery then 3.5 ml of bupivacaine 0.5% and 0.25 ml of normal saline intrathecal.

Group {M} will receive 5 ml of subcutaneous lidocaine 1% then 3.5 ml of bupivacaine 0.5% and 0.1 mg of morphine in 0.25 ml of normal saline intrathecal.

* Study procedure and anaesthetic technique
* On the arrival of patients in the operating room, an 18 gauge intravenous cannula will be inserted, and normal saline (10 ml/kg) will be infused as a preload. The patients will be connected to a monitor to record heart rate (HR), non-invasive measurement of systolic blood pressure (SBP), diastolic blood pressure (DBP), main blood pressure, continuous electrocardiogram monitoring (ECG) and oxygen saturation (SpO2). Base line reading will be recorded.
* All backup measures and equipment for general anesthesia will be ready for urgent use or rescue general anesthesia could be required.
* In the ESPB group, an ultrasound-guided ESPB will be performed on the ipsilateral side of the surgery while the patient is in lateral position using a linear 6-13 MHz ultrasound probe (SONOSITE Fujif¬ilm S-Nerve, USA) vertical parallel and 3-5 cm from the midline (10). Moving cephalic from the sacrum, we will identify the L5, L4, and L3 transverse processes and erector spinae muscles posteriorly. A 21 G and 70mm length needle (SonoPlex®, Pajunk Medizintechnologie, Germany) will be directed in-plane, and the needle tip will be positioned anterior to the erector spinae muscle at the corner of the transverse process. After the initial saline injection, dissec¬tion of the plane will be observed by injecting a total vol¬ume of 20 ml composed of 10 micrograms dexmedetomidine in 2ml of normal saline and 18 ml of bupivacaine 0.25%, which is far from the toxic dose (10). Correct placement is defined as the spread of local anesthetic cranially and caudally from the injection point, dissect¬ing the plane between the transverse processes and erector spinae muscles.
* In the intrathecal morphine group, patients will be injected with 5 ml of lidocaine subcutaneously as a local anesthetic before spinal anesthesia but using the same technique of ESPB regarding position and ultrasound guidance to ensure complete blinding of the patients.
* Patients from both groups will then receive spinal anaesthesia; intrathecal 3.5 ml hyper¬baric bupivacaine 0.5% and 0.25 ml normal saline for the E group or 0.1 mg morphine in 0.25 ml normal saline for the M group will be administered using a 25-G spinal needle inserted into the L3-L4 space with the patient in the sitting position with complete sterilization. Then patients from both groups will be allowed to be in the supine position. Sensory block will be assessed using a pin prick every 2 minutes while the patient is in the supine position until the proper level will be reached (T10 dermatome), and the Bromage scale will be measured to reach bromage 3 before surgery (11). Any decrease in heart rate below 60/min will be treated with intravenous atropine (0.01 mg/kg), and any decrease in mean arterial pressure below 20% of the basal reading will be treated by fluid bolus and 5 mg intravenous increments of ephedrine.
* Failure of ESPB technique: Technique failure will be defined as if the correct spread of local anesthetic cranially and caudally from the injection point, dissect¬ing the plane between the transverse processes and erector spinae muscles is not im¬mediately visualized (10). Those patients were not included in our study and will be replaced by other patients.
* Failure of spinal anesthesia: Technique failure will be defined as if the T10 sensory level and/or Bromage 3 scale are not reached after 20 min. of spinal injection (11). So rescue general anesthesia will be initiated; those patients not included in our study will be replaced by others.
* For both groups, oral paracetamol 1 gm./6 hours and sustained-release diclofenac 75 mg/12 hours will be administered postoperatively regularly until hospital discharge.
* IF any patient enrolled in our study complains of a pain score > 3 with regard to NPS in spite of the previously mentioned protocol for pain management, a rescue of 0.07 mg/kg IV morphine sulphate will be administrated, then NPS will be reassessed 15 minutes later if it is still > 3 a rescue 0.05 mg/kg IV morphine sulphate will be administered, which can be repeated any time postoperatively until NRS is 3 or less, provided that total morphine consumption does not exceed 0.2 mg/kg/4 hours (12).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 60 yrs. old.
* Both genders.
* ASA I, II.
* Body mass index between 20 to 30 kg per meter square.
* Height between 160 cm and 180 cm

Exclusion Criteria:

* Patient refusal.
* Age below 18 and above 60 yrs. old.
* Uncooperative patients.
* Known Allergy to the drugs enrolled in the study.
* Body mass index <30 or < 20 kg per square meter
* Any contraindication of spinal anaesthesia
* ASA III, IV patients.
* Emergency surgery.
* Neuromuscular disorder interferes with sensations in the lower limbs.
* Drug abuse or using any drug that modifies pain perception.
* Any disability affecting walking capacity rather than the operating joint.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
walking after the operation | ,patients will be allowed to walk without support at 6, 12, 18, and 24 hours postoperatively.
  Time of the first successful trial for walking 10 steps without support

SECONDARY OUTCOMES:
Postoperative pain score | 24 hours postoperative
  Postoperative pain score at 2, 4, 8, 12, and 24 hours.
Duration of hospital stay after surgery. | one week postoperative
  Duration of hospital stay after surgery.
Overall patient satisfaction with pain control. | the first 24 hours postoperatively
  • The post-operative pain score and acute postoperative pain within the first 24 hours postoperatively will be assessed using the NRS (0-10), where 0 = no pain and 10 = worst pain, at 2, 4, 8, 12, and 24 hours postoperatively.
Time of first rescue | 24 hours postopertive
  Time of first rescue: 0.07 mg/kg of morphine required by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Cairo University, Cairo, Egypt